CLINICAL TRIAL: NCT01337518
Title: A Phase 1a/1b, Open-Label Study Evaluating the Safety and Tolerability of EZN-4176, an Androgen Receptor mRNA Antagonist, in Adult Patients With Castration-Resistant Prostate Cancer
Brief Title: A Phase 1a/1b Study to Evaluate the Safety of EZN-4176, in Adult Patients With Castration-Resistant Prostate Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Reassessment of strategic direction
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZN-4176-01
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-09

CONDITIONS: Prostatic Neoplasm
Keywords: Prostate Specific Antigen; Castration Resistant Prostate Cancer; Adenocarcinoma; Androgen Receptor; Metastases
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Bulbo-Spinal Atrophy, X-Linked; Neoplasm Metastasis | interventions — 5'-ACCaagtttcttcAGC-3'

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EZN-4176 (Experimental)
  Interventions: Drug: EZN-4176

INTERVENTIONS:
Drug: EZN-4176 — EZN-4176 can be administered as a weekly one-hour i.v. infusion; weekly for 3 weeks followed by a 1 week rest; or 1 out of 2 weeks (every other week)
  Other Names: Androgen Receptor mRNA Antagonist

SUMMARY:
This study will evaluate an experimental drug called EZN-4176 to determine the anticancer effects when it is given to patients with an advanced form of prostate cancer called castration-resistant prostate cancer (CRPC). Goals of this phase I study include finding out the dose of EZN-4176 that can be safely given without serious side effects and to determine the amount of EZN-4176 that should be given in future studies.

DETAILED DESCRIPTION:
This study will be conducted in two phases:

* Phase 1a will involve dose escalation to determine the maximum tolerated dose (MTD). The MTD will be determined on the basis of the results from the safety evaluation.
* Phase 1b will involve cohort expansion at one or more dose levels to determine the recommended Phase 2 dose. The recommended Phase 2 dose, which may differ from the MTD, will be determined on the basis of results from safety, activity, and pharmacologic and correlative studies.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding protocol requirements & risks & providing written informed consent
2. Histologically or cytologically confirmed diagnosis of metastatic prostate adenocarcinoma
3. Ongoing gonadal androgen-deprivation therapy with LHRH analogs or orchiectomy. Patients without orchiectomy must receive effective LHRH analog therapy during the study
4. Testosterone < 50 ng/dL
5. Progressive disease after androgen deprivation - with all 3 of the following criteria:PSA evidence of progressive prostate cancer; PSA ≥ 5 ng/mL increasing on at least 2 successive occasions, at least 2 weeks apart. If confirmatory PSA < screening PSA, additional test for increasing PSA is needed
6. Patients receiving anti-androgen agent as part of primary androgen ablation: disease progression after stopping the anti-androgen agent. This disease progression is defined: 2 consecutive increasing PSAs ≥ 2 weeks apart, or documented osseous or soft tissue progression. Flutamide patients: at least one of the PSAs ≥ 4 weeks after stopping flutamide. Bicalutamide or nilutamide patients: at least one PSA ≥ 6 weeks after stopping the anti-androgen agent.
7. Patients who failed standard therapy or who, after physician discussion, wish to delay chemotherapy
8. Age ≥ 18 yrs
9. ECOG Score: 0-1
10. Albumin ≥3.0 g/dL
11. ANC ≥ 1,500/µL
12. Plts ≥ 75,000/µL
13. Hgb ≥ 9.0 g/dL
14. Serum Creat. ≤ 1.5xULN or Calc Creat. clearance ≥ 60 mL/min
15. Tot bili ≤ 1.5xULN
16. AST; ALT: ≤ 2.5xULN

Exclusion Criteria:

1. Prostate cancer other than adenocarcinoma, eg. neuroendocrine or small cell histology
2. Concurrent serious medical illness that might interfere with protocol compliance
3. Known chronic infectious disease, eg. AIDS or hepatitis
4. Male patient of reproductive capacity unwilling to use methods appropriate to prevent pregnancy. In the UK, double-barrier contraception required. Patients should continue to use contraception for 3 months after stopping EZN-4176 due to potential for prolonged half-life of EZN-4176 in the liver.
5. History of CNS tumor involvement
6. Other hormonal therapy, eg. megestrol acetate (Megace®), finasteride (Proscar®), dutasteride (Avodart®), or any herbal product known to decrease PSA (e.g., saw palmetto, PC-SPES, and PC-HOPE)
7. > 10 mg/day of prednisone or equivalent systemic corticosteroid within 4 weeks of first dose of EZN-4176
8. Initiation of bisphosphonates within 4 weeks of enrollment. Patients receiving stable doses of bisphosphonates with subsequent tumor progression may continue to receive this medication; however, initiation of bisphosphonates is not allowed during the study.
9. Therapy with supplements or complementary medicines/botanicals within 4 weeks of first dose of study drug, except for any combination of the following: Conventional multivitamin supplements; Selenium; Lycopene; and Soy supplements
10. Prior chemotherapy, immunotherapy, investigational therapeutic agent, or other therapy used to treat the cancer within 4 weeks (6 weeks for prior treatment with mitomycin C or nitrosoureas) before first dose of EZN-4176
11. Radiation or radioactive treatment within 4 weeks before first dose of EZN-4176. Single-fraction palliative radiation is allowed within 2 weeks before first dose of EZN-4176
12. Lack of recovery from any reversible side effects (except alopecia and Grade 1 or 2 neuropathy) to Grade 0 or 1 toxicity related to administration of an investigational therapeutic agent, chemotherapy, immunotherapy, radiotherapy, or other agents previously used to treat the cancer
13. Current participation in another clinical study with an investigational therapeutic agent and/or use of an investigational therapeutic drug (not including investigational use of an approved drug) in the 30 days before first dose of EZN-4176
14. Inability to comply with study protocol
15. Full anticoagulation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose (MTD) of EZN-4176 administered as a weekly 1-hour IV infusion. | 2012
  Evaluate incidence, severity and duration of adverse events using National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], Version 4.0, during first cycle.

SECONDARY OUTCOMES:
Determine the recommended Phase 2 dose of EZN-4176 | 2013
  Incidence, severity and duration of adverse events using National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], Version 4.0, during all cycles; Objective response, as assessed per recommendations of the Prostate Cancer Clinical Trials Working Group (PCWG2).

CONTACTS AND LOCATIONS:
Overall Officials: Aby Buchbinder, MD, Study Director — Enzon Pharmaceuticals, Inc.; Daniel Danila, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Johann de Bono, MD, Principal Investigator — Institute of Cancer Research, Royal Marsden Hospital
Locations (2):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States
- Institute of Cancer Research, Royal Marsden Hospital, Sutton, Surrey, United Kingdom